CLINICAL TRIAL: NCT00624884
Title: Velocity Vector Imaging in Patients With Moderate-to-Severe Aortic Regurgitation
Status: Completed | Type: Observational
Sponsor: Florence Nightingale Hospital, Istanbul (Other)
Responsible Party: Prof.Dr.Saide Aytekin, T.C. Istanbul Bilim University, Florence Nightingale Hospital
Other Study IDs: YT1977
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2008-06

CONDITIONS: Aortic Regurgitation
Keywords: Aortic regurgitation,velocity vector imaging
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: Patients with moderate-to-severe aortic regurgitation having normal left ventricular ejection fraction
- B: Age, sex and bodymass index matched healthy subjects

SUMMARY:
Velocity Vector Imaging may provide reliable and detailed information on left ventricular segmental function in asymptomatic patients with moderate-to severe AR. This may help to identify subclinical myocardial dysfunction in order to operate early enough to prevent postoperative heart failure and restrict unnecessary early operation which could be associated with operative risks and mortality related to prosthetic valves.

DETAILED DESCRIPTION:
Chronic aortic regurgitation (AR) is a progressive process which causes both left ventricular volume and pressure overload. While the volume overload is associated with the degree of the aortic regurgitant volume, the pressure overload occurs as a result of systemic hypertension developed due to increased stroke volume. In early stages, excentric hypertrophy occurs aiming to compensate the volume overload in the left ventricle. Therefore , ejection fraction remains in normal range despite the increasing volume overload. Left ventricular dilatation and impairment in ejection fraction only occur in the end stages of the disease. Asymptomatic patients with chronic aortic regurgitation (AR) have a good prognosis in the presence of preserved systolic function. Therefore it is a challenge to identify patients with subclinical left ventricular (LV) dysfunction. Velocity vector imaging (VVI) is a new echocardiographic method based on two dimensional gray scale imaging, which is angle independent and can provide more accurate data about cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe aortic regurgitation identified by Standard echocardiography.
* Chronic isolated aortic regurgitation
* Being asymptomatic ( Class 1 according to NYHA)
* Sinusal rhythm

Exclusion Criteria:

* Ejection fraction < 50%
* Mitral valve disease accompanied to aortic regurgitation (patients with over mild degree of mitral regurgitation and stenosis
* Aortic stenosis
* Previous myocardial infarction, or the patients with >50% coronary occlusion in any of the coronary arteries.
* Cardiomyopathies
* AV conduction disorders
* Chronic renal or hepatic insufficiency
* Malignities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tertiary care clinic
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Velocity Vector Imaging derived segmental systolic peak Strain and Strain rates | April 2008

CONTACTS AND LOCATIONS:
Overall Officials: Saide Aytekin, Professor, Principal Investigator — T.C. Istanbul Bilim University, Florence Nightingale Hospital, Division of Cardiology
Locations (1):
- TC.Istanbul Bilim University, Florence Nightingale Hospital, Division of Cardiology, Istanbul, Sisli, Turkey (Türkiye)

REFERENCES:
- [Background] Sokmen G, Sokmen A, Duzenli A, Soylu A, Ozdemir K. Assessment of myocardial velocities and global function of the left ventricle in asymptomatic patients with moderate-to-severe chronic aortic regurgitation: a tissue Doppler echocardiographic study. Echocardiography. 2007 Jul;24(6):609-14. doi: 10.1111/j.1540-8175.2007.00438.x. PMID 17584200